CLINICAL TRIAL: NCT01626469
Title: Eye Blood Flow and the Kidney
Brief Title: Measurement of Eye Blood Flow and Renal Function in Healthy and Diabetic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Norman K. Hollenberg, MD, PhD, Director of Physiologic Research Division, Department of Radiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011P002805
Record Dates: First submitted 2012-06-19; First posted 2012-06-22 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Captopril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Captopril 25 mg (Admission 1, Day 1, low salt diet) Matched Placebo (Admission 1, Day 2, low salt diet) Captopril 25 mg (Admission 2, Day 1, high salt diet) Matched Placebo (Admission 2, Day 2, high salt diet)
  Interventions: Drug: Captopril; Drug: placebo
- Captopril (Placebo Comparator): Matched Placebo (Admission 1, Day 1, low salt diet) Captopril 25 mg (Admission 1, Day 2, low salt diet) Matched Placebo (Admission 2, Day 1, high salt diet) Captopril 25 mg (Admission 2, Day 2, high salt diet)
  Interventions: Drug: Captopril; Drug: placebo

INTERVENTIONS:
Drug: Captopril — 25mg Captopril
Drug: placebo — placebo

SUMMARY:
The purpose of this study is to the determine the effect of salt intake and Captopril on the ophthalmic artery (OA) blood supply of individuals with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
The overall objective of this study is to ascertain if salt intake affects ophthalmic artery (OA) blood flow. In addition, we will study both the eye and kidney response to ACE inhibition compared to placebo while controlling salt intake in subjects with Type 2 diabetes mellitus.

We hypothesize that salt intake will affect OA blood flow.

We will initially look at both eye and renal response to subjects on a low salt diet (10mEq Na/day) followed by response to high salt diet (200mEq Na/day). In addition, we may look at eye response while subjects consume their regular diet.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Heart Attack or Stroke within the last 6 months
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in ophthalmic artery blood flow from baseline | 1 hour post drug, 2 hours post drug, 3 hours post drug
  Eye blood flow will be measured at baseline and post drug time points (3 total)

SECONDARY OUTCOMES:
Change in blood pressure from baseline | Every 15 minutes for 3 hours
  Blood pressure will be monitored throughout the study starting at baseline
Change in renal plasma flow (RPF) from baseline | 1 hour post drug, 2 hours post drug, 3 hours post drug
  Renal Plasma Flow (to measure kidney function) will be measured at baseline and post drug time points (3 total)

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Hollenberg, MD, PhD, Principal Investigator — Brigham and Women's Hospital; Ebrahim Barkoudah, M.D.,M.P.H., Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States